CLINICAL TRIAL: NCT00462475
Title: Phase 4 Study of Recombinant GH on Intima-Media Thickness at Common Carotids and on Cardiovascular Risk Factors in Hypopituitary Patients
Brief Title: Effect of 5 Years of GH Replacement on Atherosclerosis
Acronym: 5yrGH
Status: Completed | Type: Observational
Sponsor: Federico II University (Other)
Other Study IDs: NeuroendoUnit-3
Record Dates: First submitted 2007-04-18; First posted 2007-04-19 (Estimated); Last update posted 2007-10-16 (Estimated); Status verified 2007-10

CONDITIONS: Hypopituitarism; Pituitary Tumors; Growth Hormone Deficiency
Keywords: GH; IGF-I; GH deficiency; Atherosclerosis; Insulin resistance syndrome
MeSH Terms: conditions — Hypopituitarism; Pituitary Neoplasms; Dwarfism, Pituitary; Atherosclerosis; Metabolic Syndrome | interventions — Growth Hormone; Human Growth Hormone

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Recombinant Growth Hormone, Genotropin (Pfizer)

SUMMARY:
Adult patients with hypopituitarism under adequate conventional hormone replacement therapy have reduced life expectancy due to excess vascular events (1-4). Deficiency in GH secretion (GHD) is likely to play a major role in determining the excess mortality, since it is associated with lipid abnormalities, visceral adiposity, glucose intolerance, insulin resistance, hypertension, cardiac abnormalities and increased intima-media thickness (IMT) at major arteries (5).

Beneficial effects of growth hormone (GH) replacement on cardiovascular risk factors have been demonstrated in several studies of hypopituitary GHD patients (5). GH replacement improves body composition and lipid profile (5): it is accepted that management of dyslipidaemia is crucial in primary and secondary prevention of cardiovascular disease and part of the excess vascular risk associated with hypopituitarism is likely to be due to dyslipidaemia (6). A meta-analysis of blinded, randomized, placebo-controlled trials with low doses and long-duration GH treatment showed that GH replacement has beneficial effects on cardiovascular risk by improving lean and fat body mass, total and LDL cholesterol levels, and diastolic blood pressure (7). Besides, GH replacement also induces improvement in cardiovascular markers (8), and cardiac performance (9). In small cohorts of GHD adults, beneficial effects of GH replacement for 6-24 mos have also been reported on surrogate parameters of atherosclerosis, such as intima-media thickness (IMT) at major arteries (10-13), while 6 months of GH deprivation is associated with an impairment of the cardiovascular risk profile (12). In a consistent series of men and women with hypopituitarism we reported, however, that two years of GH replacement is not adequate to normalize IMT levels at common carotid arteries (13).

To give further insights on the likelihood of reversal of early atherosclerosis in severe GHD patients after prolonged GH replacement, we designed this 5-yr prospective, controlled study. Only men aged ≤50 yrs and with severe GHD were enrolled to avoid gender and aging interference (13). Main outcome measure was IMT at common carotid arteries; secondary measure was prevalence of insulin-resistance syndrome according with the American College of Endocrinology (14).

DETAILED DESCRIPTION:
This is an observational,5-yr prospective, controlled study. At study entry, all subjects underwent serum assay of IGF-I, systolic and diastolic blood pressure (SBP, DBP) measurement, total-, and HDL-cholesterol, triglycerides, glucose, and insulin level after an overnight fasting, and common carotid arteries ultrasonography. The oral glucose load (oGTT) was performed by measuring blood glucose every 30 minutes for 2 hours after the oral administration of 75 g of glucose diluted in 250 ml of saline solution. The conversion factors (mg/dl to mmol/l) for lipids and glucose were as follows: cholesterol 0.02586, triglycerides 0.01129, and glucose 0.05551. According with previous studies (13,19-21) blood pressure was measured at the right arm, with the subjects in relaxed sitting position. The average of six measurements (three taken by each of two examiners, in the same day, between 8.00-9.00 in the morning) with a mercury sphygmomanometer was used in all analysis.

In the patients, all parameters and carotid ultrasonography were re-evaluated after 12, 24, 36, 48 and 60 months while in controls they were re-evaluated after 60 months.

At study entry and at study end, in all of the patients and controls the prevalence of insulin-resistance syndrome (IRS) was evaluated according with the American College of Endocrinology (14) based on the presence of at least two criteria of the following: triglycerides levels ≥1.7 mmol/liter, HDL-cholesterol levels ≤1.0 mmol/liter, blood pressure above 130/85 mmHg, fasting glucose between 6.1 and 7 mmol/liter or 2 hr after oGTT between 7.7 and 11.1 mmol/liter.

ELIGIBILITY:
Inclusion Criteria:

* male gender
* age <50 yrs to limit the effect of aging;
* body mass index <30 Kg/m2;
* no familial or personal history of cardiovascular diseases;
* no concomitant treatment with drugs known to interfere with glucose or lipid metabolism or to influence blood pressure at the time of study entry;
* no previous GH treatment

Exclusion Criteria:

* female gender
* age >50 yrs;
* body mass index ≥30;
* familial or personal history of cardiovascular diseases;
* previous and present treatments with drugs known to interfere with glucose or lipid metabolism or to influence blood pressure;
* previous GH treatment in adult age
* GHD of childhood onset
* GHD due to previous Cushing's disease

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Three groups are studied: 1) Males with severe GHD undergoing GH replacement; 2) Males with severe GHD who did not undergo GH replacement because of either refusal or presence of risk factors for this treatment; 2) control men, age-matched with the patients.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 1996-01; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Intima-media thickness at common carotid arteries at baseline and after 5 years | 5 yrs

SECONDARY OUTCOMES:
Prevalence of insulin resistance (IR) syndrome (IRS) and LDL/HDL-cholesterol ratio at baseline and after 5 years | 5 yrs

CONTACTS AND LOCATIONS:
Overall Officials: Annamaria AL Colao, Prof., Principal Investigator — University "Federico II"
Locations (1):
- Department of Molecular and Clinical Endocirnology and Oncology University Federico II of Naples, Naples, Italy

REFERENCES:
- [Result] Rosen T, Bengtsson BA. Premature mortality due to cardiovascular disease in hypopituitarism. Lancet. 1990 Aug 4;336(8710):285-8. doi: 10.1016/0140-6736(90)91812-o. PMID 1973979
- [Result] Bulow B, Hagmar L, Mikoczy Z, Nordstrom CH, Erfurth EM. Increased cerebrovascular mortality in patients with hypopituitarism. Clin Endocrinol (Oxf). 1997 Jan;46(1):75-81. doi: 10.1046/j.1365-2265.1997.d01-1749.x. PMID 9059561
- [Result] Bates AS, Van't Hoff W, Jones PJ, Clayton RN. The effect of hypopituitarism on life expectancy. J Clin Endocrinol Metab. 1996 Mar;81(3):1169-72. doi: 10.1210/jcem.81.3.8772595.
- [Result] Tomlinson JW, Holden N, Hills RK, Wheatley K, Clayton RN, Bates AS, Sheppard MC, Stewart PM. Association between premature mortality and hypopituitarism. West Midlands Prospective Hypopituitary Study Group. Lancet. 2001 Feb 10;357(9254):425-31. doi: 10.1016/s0140-6736(00)04006-x. PMID 11273062
- [Result] Colao A, Di Somma C, Savanelli MC, De Leo M, Lombardi G. Beginning to end: cardiovascular implications of growth hormone (GH) deficiency and GH therapy. Growth Horm IGF Res. 2006 Jul;16 Suppl A:S41-8. doi: 10.1016/j.ghir.2006.03.006. Epub 2006 May 11. PMID 16690338
- [Result] Abdu TA, Neary R, Elhadd TA, Akber M, Clayton RN. Coronary risk in growth hormone deficient hypopituitary adults: increased predicted risk is due largely to lipid profile abnormalities. Clin Endocrinol (Oxf). 2001 Aug;55(2):209-16. doi: 10.1046/j.1365-2265.2001.01320.x. PMID 11531927
- [Result] Maison P, Griffin S, Nicoue-Beglah M, Haddad N, Balkau B, Chanson P; Metaanalysis of Blinded, Randomized, Placebo-Controlled Trials. Impact of growth hormone (GH) treatment on cardiovascular risk factors in GH-deficient adults: a Metaanalysis of Blinded, Randomized, Placebo-Controlled Trials. J Clin Endocrinol Metab. 2004 May;89(5):2192-9. doi: 10.1210/jc.2003-030840. PMID 15126541
- [Result] Gola M, Bonadonna S, Doga M, Giustina A. Clinical review: Growth hormone and cardiovascular risk factors. J Clin Endocrinol Metab. 2005 Mar;90(3):1864-70. doi: 10.1210/jc.2004-0545. Epub 2004 Dec 7. PMID 15585563
- [Result] Colao A, Marzullo P, Di Somma C, Lombardi G. Growth hormone and the heart. Clin Endocrinol (Oxf). 2001 Feb;54(2):137-54. doi: 10.1046/j.1365-2265.2001.01218.x. PMID 11207626
- [Result] Pfeifer M, Verhovec R, Zizek B, Prezelj J, Poredos P, Clayton RN. Growth hormone (GH) treatment reverses early atherosclerotic changes in GH-deficient adults. J Clin Endocrinol Metab. 1999 Feb;84(2):453-7. doi: 10.1210/jcem.84.2.5456. PMID 10022400
- [Result] Borson-Chazot F, Serusclat A, Kalfallah Y, Ducottet X, Sassolas G, Bernard S, Labrousse F, Pastene J, Sassolas A, Roux Y, Berthezene F. Decrease in carotid intima-media thickness after one year growth hormone (GH) treatment in adults with GH deficiency. J Clin Endocrinol Metab. 1999 Apr;84(4):1329-33. doi: 10.1210/jcem.84.4.5595. PMID 10199774
- [Result] Colao A, Di Somma C, Rota F, Pivonello R, Savanelli MC, Spiezia S, Lombardi G. Short-term effects of growth hormone (GH) treatment or deprivation on cardiovascular risk parameters and intima-media thickness at carotid arteries in patients with severe GH deficiency. J Clin Endocrinol Metab. 2005 Apr;90(4):2056-62. doi: 10.1210/jc.2004-2247. Epub 2005 Jan 25. PMID 15671089
- [Result] Colao A, Di Somma C, Cuocolo A, Spinelli L, Acampa W, Spiezia S, Rota F, Savanelli MC, Lombardi G. Does a gender-related effect of growth hormone (GH) replacement exist on cardiovascular risk factors, cardiac morphology, and performance and atherosclerosis? Results of a two-year open, prospective study in young adult men and women with severe GH deficiency. J Clin Endocrinol Metab. 2005 Sep;90(9):5146-55. doi: 10.1210/jc.2005-0597. Epub 2005 Jun 28. PMID 15985481
- [Result] Einhorn D, Reaven GM, Cobin RH, Ford E, Ganda OP, Handelsman Y, Hellman R, Jellinger PS, Kendall D, Krauss RM, Neufeld ND, Petak SM, Rodbard HW, Seibel JA, Smith DA, Wilson PW. American College of Endocrinology position statement on the insulin resistance syndrome. Endocr Pract. 2003 May-Jun;9(3):237-52. No abstract available. PMID 12924350
- [Result] Aimaretti G, Corneli G, Razzore P, Bellone S, Baffoni C, Arvat E, Camanni F, Ghigo E. Comparison between insulin-induced hypoglycemia and growth hormone (GH)-releasing hormone + arginine as provocative tests for the diagnosis of GH deficiency in adults. J Clin Endocrinol Metab. 1998 May;83(5):1615-8. doi: 10.1210/jcem.83.5.4837. PMID 9589665
- [Result] Colao A, Di Somma C, Filippella M, Rota F, Pivonello R, Orio F, Vitale G, Lombardi G. Insulin-like growth factor-1 deficiency determines increased intima-media thickness at common carotid arteries in adult patients with growth hormone deficiency. Clin Endocrinol (Oxf). 2004 Sep;61(3):360-6. doi: 10.1111/j.1365-2265.2004.02105.x. PMID 15355453
- [Result] Colao A, Cerbone G, Pivonello R, Aimaretti G, Loche S, Di Somma C, Faggiano A, Corneli G, Ghigo E, Lombardi G. The growth hormone (GH) response to the arginine plus GH-releasing hormone test is correlated to the severity of lipid profile abnormalities in adult patients with GH deficiency. J Clin Endocrinol Metab. 1999 Apr;84(4):1277-82. doi: 10.1210/jcem.84.4.5605. PMID 10199767
- [Result] Colao A, Di Somma C, Pivonello R, Loche S, Aimaretti G, Cerbone G, Faggiano A, Corneli G, Ghigo E, Lombardi G. Bone loss is correlated to the severity of growth hormone deficiency in adult patients with hypopituitarism. J Clin Endocrinol Metab. 1999 Jun;84(6):1919-24. doi: 10.1210/jcem.84.6.5742. PMID 10372687
- [Result] Colao A, Di Somma C, Cuocolo A, Filippella M, Rota F, Acampa W, Savastano S, Salvatore M, Lombardi G. The severity of growth hormone deficiency correlates with the severity of cardiac impairment in 100 adult patients with hypopituitarism: an observational, case-control study. J Clin Endocrinol Metab. 2004 Dec;89(12):5998-6004. doi: 10.1210/jc.2004-1042. PMID 15579750
- [Result] Colao A, di Somma C, Cuocolo A, Spinelli L, Tedesco N, Pivonello R, Bonaduce D, Salvatore M, Lombardi G. Improved cardiovascular risk factors and cardiac performance after 12 months of growth hormone (GH) replacement in young adult patients with GH deficiency. J Clin Endocrinol Metab. 2001 May;86(5):1874-81. doi: 10.1210/jcem.86.5.7464. PMID 11344175
- [Result] Colao A, di Somma C, Pivonello R, Cuocolo A, Spinelli L, Bonaduce D, Salvatore M, Lombardi G. The cardiovascular risk of adult GH deficiency (GHD) improved after GH replacement and worsened in untreated GHD: a 12-month prospective study. J Clin Endocrinol Metab. 2002 Mar;87(3):1088-93. doi: 10.1210/jcem.87.3.8336. PMID 11889170
- [Derived] Colao A, Di Somma C, Spiezia S, Savastano S, Rota F, Savanelli MC, Lombardi G. Growth hormone treatment on atherosclerosis: results of a 5-year open, prospective, controlled study in male patients with severe growth hormone deficiency. J Clin Endocrinol Metab. 2008 Sep;93(9):3416-24. doi: 10.1210/jc.2007-2810. Epub 2008 Jul 1. PMID 18593773